CLINICAL TRIAL: NCT03403504
Title: An Open-label, Single Dose, Randomised, Cross-over Study to Determine the Fasted State Pharmacokinetics of Oxycodone From Oxycodone Tamper Resistant (OTR) Tablet 10 mg and OXYCONTIN® Tablet 10 mg in Chinese Subjects With Chronic Pain
Brief Title: OTR Tablet 10 mg Fasted-state Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ONF16-CN-101
Record Dates: First submitted 2016-07-26; First posted 2018-01-18 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Receptors, Oxytocin; Tablets; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone Tamper Resistant (Experimental): Oxycodone Tamper Resistant (OTR) Tablet 10 mg
  Interventions: Drug: Oxycodone Tamper Resistant
- OXYCONTIN® (Active Comparator): OXYCONTIN® Tablet 10 mg
  Interventions: Drug: OXYCONTIN®

INTERVENTIONS:
Drug: Oxycodone Tamper Resistant — Orally administered Oxycodone Tamper Resistant 10mg
  Other Names: Oxycodone Tamper Resistant (OTR) Tablet 10 mg
  Arms: Oxycodone Tamper Resistant
Drug: OXYCONTIN® — Orally administered OXYCONTIN® Tablet 10 mg
  Other Names: OXYCONTIN® Tablet 10 mg
  Arms: OXYCONTIN®

SUMMARY:
This is an open-label, single Dose, randomised, cross-over study to confirm the bioequivalence (BE) of OTR tablet 10 mg and OXYCONTIN tablet 10 mg in a fasted state in Chinese subjects with chronic pain

DETAILED DESCRIPTION:
The investigation is designed as an open-label, single dose, randomized, and cross-over study to determine the PK profile of oxycodone from OTR tablet 10 mg and OXYCONTIN tablet 10 mg in Chinese subjects with chronic pain in a fasted state.

the China regulations for drug registration require that controlled medicine (opioid is categorized to be a controlled medicine) should not be applied in healthy volunteers in clinical studies. In this BE study, subjects with histories of chronic pain are chosen as the target population.

Inclusion/exclusion criteria are strictly defined to reduce the potential variation of the PK data. The subjects with abnormal liver and kidney functions, which may affect the metabolism of oxycodone.

As a general rule, cross-over design is applied in the study to decrease the inter-individual variations between the two cohorts. A washout period lasting for at least 7 half-lives of the investigational medicine is needed to eliminate the drug residual from the previous period

open label design is applied since the plasma concentration of oxycodone is to be objectively tested and analysed and randomization will be applied to reduce selection bias.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female subjects with histories of chronic pain regardless of the aetiology, aged 18-55 years both inclusive
2. The average pain over the last 24 hours should be scored < 4 assessed with Numeric Rating Scales (NRS), when not receiving analgesics. The pain condition has been kept stable at least in the past 7 days prior to entering into the screening and is expected to be stable during the study duration
3. Body weight ≥45 kg and a body mass index (BMI) ≥18 and ≤28 kg/m2
4. Karnofsky score of Performance Status ≥70
5. Willing to take all the food supplied while the subject is in the study unit
6. Be able to read, understand, and sign written Informed Consent Form (ICF) prior to study participation and be willing to follow the protocol requirements
7. Willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, some Intrauterine Device (IUD), sexual abstinence, or vasectomised partner
8. Female subjects, including those up to less than one year post-menopausal, must have a negative serum pregnancy test and be non-lactating.

Exclusion Criteria:

1. Subjects who are currently taking opioids or have used opioids in the past 14 days prior to receiving the study drug
2. Have hypersensitivity history to any opioids, naltrexone, naloxone, or related compounds or any contraindications as detailed in the OTR and OXYCONTIN tablet Summary of Product Characteristics
3. Histories of or any current conditions that might interfere with drug absorption, distribution, metabolism, or excretion
4. Subjects who are likely to have paralytic ileus or acute abdomen or to require an operation on abdominal regions
5. Subjects with biliary tract diseases, pancreatitis, prostatic hypertrophy, or corticoadrenal insufficiency
6. Subjects with respiratory depression, corpulmonale, or chronic bronchial asthma
7. Any history of seizures or symptomatic head trauma
8. Subjects with abnormal liver function (values exceeding the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin during the Screening Phase) or abnormal renal function (values exceeding the ULN for serum creatinine during the Screening Phase). Note: if the values of ALT, AST or total bilirubin are between 1 to 1.2 times of ULN and confirmed not clinically significant by the Investigators, the subject may be recruited after getting the approval from Sponsor.
9. Any other significant illness other than the primary disease of chronic pain during the 4 weeks preceding the entry into this study
10. Subjects who are unable to stop taking monoamine oxidase inhibitors during this trial period or time lapses less than 2 weeks since drug withdrawal prior to the study drug administration
11. Subjects who are currently taking tricyclic antidepressants or have used tricyclic antidepressants within 4 weeks prior to the study drug administration
12. Subjects who have used any medicinal product which inhibits Cytochrome P450 3A4 (CYP3A4) (e.g. troleandomycin, ketoconazole, gestodene, etc.) or induces CYP3A4 (e.g. glucocorticoids, barbiturates, rifampicin, etc.) within 4 weeks prior to the study drug administration
13. Subjects who have used any medicinal product which inhibits Cytochrome P450 2D6 (CYP2D6) (e.g. fluoxetine, quinidine, ritonavir, etc.) or induces CYP2D6 (e.g. dexamethasone, rifampicin, glutethimide, etc.) within 4 weeks prior to the study drug administration
14. Histories of smoking (being a smoker or an occasional smoker) within 45 days prior to the study drug administration and refusal to abstain from smoking during the study. According to World Health Organization (WHO), a smoker is defined as having smoked at least 1 cigarette per day continuously for more than 6 months and an occasional smoker is defined as having smoked for more than 4 times per week and less than 1 cigarette per day continuously for more than 6 months.
15. Subjects with histories of alcoholism or drug abuse. Alcoholism is defined as regular alcohol consumption exceeding 14 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor)
16. Consumption of alcoholic beverages within 48 hours before study drug administration, and refusal to abstain from alcohol for at least 48 hours after study drug administration
17. Refusal to abstain from food for 10 hours preceding and 4 hours following administration of the study drug and to abstain from caffeine or xanthine entirely during each confinement
18. Positive Hepatitis B Surface Antigen (HBsAg), anti-Hepatitis C Virus (HCV), anti-Human Immunodeficiency Virus (HIV), or syphilis antibody test result
19. Urine screening before study is positive for opioids, barbiturates, amphetamines, cocaine metabolites, methadone, benzodiazepines, phencyclidine, methamphetamine, or cannabinoids. Or alcohol breath test is positive
20. Any history of frequent nausea or emesis regardless of aetiology
21. Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol
22. Subjects who participated in a clinical research study within 30 days of study entry

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenping Wang, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine
Locations (1):
- The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24, from Mar2017 to Jul2017, from patient database, medical clinic, advertisement recruitment and etc.
Groups:
- OXYCONTIN 10 mg - OTR 10 mg: the treatment sequence is OXYCONTIN 10 mg dose first and then OTR 10 mg dose in fasted state
- OTR 10 Mg-OXYCONTIN 10 mg: the treatment sequence is OTR 10 mg dose first and then OXYCONTIN 10 mg dose in fasted state
Period: Period 1
Arm/Group | OXYCONTIN 10 mg - OTR 10 mg | OTR 10 Mg-OXYCONTIN 10 mg
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Period: Period 2
Arm/Group | OXYCONTIN 10 mg - OTR 10 mg | OTR 10 Mg-OXYCONTIN 10 mg
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OXYCONTIN 10 Mg-OTR 10 mg: the treatment sequence is OXYCONTIN 10 mg dose first and then OTR 10 mg dose
- OTR 10 Mg-OXYCONTIN 10 mg: the treatment sequence is OTR 10 mg dose first and then OXYCONTIN 10 mg dose
- Total: Total of all reporting groups
Arm/Group | OXYCONTIN 10 Mg-OTR 10 mg | OTR 10 Mg-OXYCONTIN 10 mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 36.9 (10.18) | 41.6 (10.44) | 39.3 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HAN | 10 | 12 | 22
  Other | 2 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 68.29 (11.462) | 64.25 (9.536) | 66.27 (10.516)
Height [Mean (Standard Deviation); unit: cm] | 169.3 (8.11) | 167.9 (5.70) | 168.6 (6.89)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.72 (2.888) | 22.76 (2.974) | 23.24 (2.908)

OUTCOME MEASURES:

1. Primary Outcome: Cmax of OTR Tablet 10 mg and OXYCONTIN Tablet 10 mg in a Fasted State
Description: The analysis was for PK parameters Cmax of analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) were used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng/ml
Groups:
- Cmax of OTR 10 mg: the treatment group with OTR 10 mg
- Cmax of OXYCONTIN 10 mg: the treatment group with OXYCONTIN 10 mg
Arm/Group | Cmax of OTR 10 mg | Cmax of OXYCONTIN 10 mg
Number analyzed (Participants) | 23 | 23
ng/ml | 11.617 [8.5821 to 14.6519] | 10.564 [8.3103 to 12.8177]

2. Primary Outcome: AUCt of OTR Tablet 10 mg and OXYCONTIN Tablet 10 mg in a Fasted State
Description: The analysis was for PK parameters AUCt of analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) were used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng*h/ml
Groups:
- AUCt of OTR Tablet 10 mg: OTR tablet 10 mg
- AUCt of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | AUCt of OTR Tablet 10 mg | AUCt of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
ng*h/ml | 123.5608 [93.4687 to 153.6529] | 124.0294 [98.1652 to 149.8936]

3. Primary Outcome: AUCINF of OTR Tablet 10 mg and OXYCONTIN Tablet 10 mg in a Fasted State
Description: The analysis was for PK parameters AUCINF for analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) was used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng*h/ml
Groups:
- AUCINF of OTR Tablet 10 mg: OTR tablet 10 mg
- AUCINF of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | AUCINF of OTR Tablet 10 mg | AUCINF of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
ng*h/ml | 125.7605 [94.4572 to 157.0638] | 127.4811 [100.0286 to 154.9336]

4. Secondary Outcome: Adverse Events of OTR Tablet 10 mg and OXYCONTIN Tablet 10 mg, When Given to Chinese Subjects With Chronic Pain in a Fasted State
Description: An overall summary of the number and percentage of Adverse Events will be provided for each treatment groups to assess the safety of OTR tablet 10 mg and OXYCONTIN tablet 10 mg.
Time Frame: up to 35 days
Measure: Number; unit: AEs
Groups:
- Adverse Events of OTR Tablet 10 mg: OTR tablet 10 mg
- Adverse Events of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | Adverse Events of OTR Tablet 10 mg | Adverse Events of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
AEs
  Number of AEs | 17 | 13
  Number of TEAEs | 17 | 13
  Number of related TEAEs | 8 | 6

5. Secondary Outcome: Number of AEs Related to Vital Signs
Description: Vital sign parameters( systolic blood pressure, diastolic blood pressure, pulse rate, respiration rate, and axillary temperature)to be summarised on the rate of lower than, within, and higher than the reference range values from baseline to end of study.
Time Frame: up to 35 days
Measure: Number; unit: AEs of vital signs related
Groups:
- Vital Signs of OTR Tablet 10 mg: OTR tablet 10 mg
- Vital Signs of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | Vital Signs of OTR Tablet 10 mg | Vital Signs of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
AEs of vital signs related | 7 | 5

6. Secondary Outcome: Number of AEs Related to ECGs
Description: Twelve-lead ECG was conducted at screening and on Day 4 of Period 2.
Time Frame: up to 35 days
Measure: Number; unit: AEs related to ECGs
Groups:
- ECG of OTR Tablet 10 mg: OTR tablet 10 mg and OXYCONTIN tablet 10 mg
- ECG of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | ECG of OTR Tablet 10 mg | ECG of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
AEs related to ECGs | 0 | 0

7. Secondary Outcome: Number of Lab Tests With Clinical Significance
Description: Clinical laboratory data (hematology, blood chemistry, and urinalysis) to be summarized on the rate of lower than, within, and higher than the reference range values from baseline to end of study.
Time Frame: up to 35 days
Measure: Number; unit: lab tests with clinical significance
Groups:
- Clinical Laboratory Data of OTR Tablet 10 mg: OTR tablet 10 mg
- Clinical Laboratory Data of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | Clinical Laboratory Data of OTR Tablet 10 mg | Clinical Laboratory Data of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
lab tests with clinical significance | 6 | 3

8. Secondary Outcome: Number of AEs Related to Physical Examination
Description: Physical examination was conducted at screening, and on Day -1, Day 4 in each Period.
Time Frame: up to 35 days
Measure: Number; unit: AEs related to physical examinations
Groups:
- Physical Examinations of OTR Tablet 10 mg: OTR tablet 10 mg
- Physical Examinations of OXYCONTIN Tablet 10 mg: OXYCONTIN tablet 10 mg
Arm/Group | Physical Examinations of OTR Tablet 10 mg | Physical Examinations of OXYCONTIN Tablet 10 mg
Number analyzed (Participants) | 23 | 23
AEs related to physical examinations | 0 | 0

ADVERSE EVENTS:
Time Frame: Events will be recorded from the point at which the ICF is signed until 7±1 days after last oxycodone dose in the case of completion/discontinuation from the study. This includes new AEs that are reported within 7±1 days after last oxycodone dosing after the subject's completion/discontinuation visit. AE data has been collected for 35 days since ICF signed up to follow-up visit for study completion of each subject.
Description: same with clinicaltrials.gov Definitions.
Groups:
- OTR 10 mg: the treatment group with OTR 10 mg
- OXYCONTIN 10 mg: the treatment group with OXYCONTIN 10 mg
Arm/Group | OTR 10 mg | OXYCONTIN 10 mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7/23 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTR 10 mg (N=23) | OXYCONTIN 10 mg (N=23)
Heart rate decreased (Cardiac disorders) | 4 (4) | 0 (0)
WBC urine positive (Renal and urinary disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03403504/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03403504/SAP_001.pdf